CLINICAL TRIAL: NCT03224936
Title: Propofolsleep - A Observational Study on Cardiopulmonary and Pharyngeal Reactions While Drug Induced Sleep Endoscopy in Patients With Obstructive Sleep Apnea Syndrome Under PSI Monitoring
Brief Title: Propofolsleep - A Study on Cardiopulmonary and Pharyngeal Reactions While Drug Induced Sleep Endoscopy (DISE)
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Treskatsch, Deputy head of department Department of Anesthesiology and Operative Intensive Care Medicine, CCM and CVK, Charite University, Berlin, Germany
Other Study IDs: Propofolschlaf
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Sleep Apnea, Obstructive; Electroencephalography; Echocardiography; Blood Gas Monitoring, Transcutaneous; Consciousness Monitors
Keywords: DISE; OSAS; PSI
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DISE group: All patients in this study group will receive a propofol PSI controlled DISE (drug induced sleep endoscopy).
  Interventions: Device: PSI

INTERVENTIONS:
Device: PSI — The PSI delivered by Masimo Root (Sedline) will be measured in all patients.

SUMMARY:
While Drug Induced Sleep Endoscopy (DISE) in patients with obstructive sleep apnea syndrome (OSAS) apnea and hypopnea occur. Because of the induced phases of apnea in a controlled setting it is possible to evaluate the related pathophysiology of apnea. We plan to correlate the Patient State Index (PSI) and other physiologic parameters with phases of apnea and hypopnea.

DETAILED DESCRIPTION:
DISE is a standard method in diagnosis of OSAS and its specific localisation and severity. 20 patients with polysomnographic diagnosed OSAS will be enrolled in this prospective observational study. All patients would get a DISE because of the before mentioned reasons (localisation and severity) although they wouldn't participate in this study. They will get a 24-h-RR (blood pressure)-measurement, a transthoracic echocardiography, a peak-flow-test and routine lab examination including troponin and proBNP before the examination. Furthermore they have to fill out the Epworth Sleepiness Scale questionaire.

Before starting the DISE a standard-monitoring (Electrocardiography, pulse oximetry, non-invasive blood pressure, patient state index, near infrared spectroscopy, transcutaneous CO2 (carbon dioxide), invasive blood pressure) will be established. After applying the monitoring the DISE is started by target controlled infusion (Marsh Model) with a sighted goal-concentration of 3.0 µg/ml Propofol in 5 minutes. While the examination a stabile snoring-phase with apnoea/hypopnoea is needed. In this moment a video-endoscopy is started to quantify the level of obstruction. After DISE the sedation will end and the patients will be transported to the recovery room or postanesthesia care unit (PACU). For specific order of events a video recording of the DISE will be realized.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent
* age of 18 years or older
* no participation in other prospective interventional studies
* OSAS with a polysomnographic shown AHI (apnea-hypopnea-index) of 15/h or more

Exclusion Criteria:

* no written informed consent
* allergies against study medication
* ASA (american society of anesthesiologists) class 4 or higher
* neurodegenerative CNS (central nerve system) or muscle diseases
* pregnant or breastfeeding patients
* 25 % or more central or mixed apneas in polysomnography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years or older voluntary patients with an obstructive sleep apnea syndrome undergoing elective propofol induced sleep endoscopy at Charité - Universitätsmedizin Berlin Campus Charite Mitte.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PSI | Duration of surgery (an average of 2 hours)
  Depth of sedation is monitored with a SEDline electroencephalograph based monitor that displays patient state index (PSI).

SECONDARY OUTCOMES:
NIRS (near-infrared spectrometry) | Duration of surgery (an average of 2 hours)
  Near-infrared spectrometry in % of left and right hemisphere
transcutaneous CO2 (carbon dioxide) | Duration of surgery (an average of 2 hours)
  Measured at the chest.
transcutaneous O2 (oxygen) | Duration of surgery (an average of 2 hours)
  Measured at the center of the chest.
Propofol | Duration of surgery (an average of 2 hours)
  Total amount of administered propofol.
Diaphragma movement | Duration of surgery (an average of 2 hours)
  Diaphragma movement is measured by ultrasound.
blood gases | Duration of surgery (an average of 2 hours)
  Arterial blood gas is obtained from an arterial line.
heart rate | Duration of surgery (an average of 2 hours)
  by ECG.
blood pressure | Duration of surgery (an average of 2 hours)
  NIBP and IBP.
TTE (transthoracic echocardiography) | shortly before DISE (an average of 30 minutes)
  Parameters of left and right ventricular function, as well as function of heart valves before DISE.
EEG parameters | Duration of surgery (an average of 2 hours)
  Parameters measured by the Sedline monitor

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Treskatsch, MD, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin Campus Charité Mitte, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franklin KA, Lindberg E. Obstructive sleep apnea is a common disorder in the population-a review on the epidemiology of sleep apnea. J Thorac Dis. 2015 Aug;7(8):1311-22. doi: 10.3978/j.issn.2072-1439.2015.06.11. PMID 26380759
- [Background] Rivas M, Ratra A, Nugent K. Obstructive sleep apnea and its effects on cardiovascular diseases: a narrative review. Anatol J Cardiol. 2015 Nov;15(11):944-50. doi: 10.5152/AnatolJCardiol.2015.6607. PMID 26574763
- [Background] Drager LF, Togeiro SM, Polotsky VY, Lorenzi-Filho G. Obstructive sleep apnea: a cardiometabolic risk in obesity and the metabolic syndrome. J Am Coll Cardiol. 2013 Aug 13;62(7):569-76. doi: 10.1016/j.jacc.2013.05.045. Epub 2013 Jun 12. PMID 23770180
- [Background] Kaneko Y, Floras JS, Usui K, Plante J, Tkacova R, Kubo T, Ando S, Bradley TD. Cardiovascular effects of continuous positive airway pressure in patients with heart failure and obstructive sleep apnea. N Engl J Med. 2003 Mar 27;348(13):1233-41. doi: 10.1056/NEJMoa022479. PMID 12660387
- [Background] Mansfield DR, Gollogly NC, Kaye DM, Richardson M, Bergin P, Naughton MT. Controlled trial of continuous positive airway pressure in obstructive sleep apnea and heart failure. Am J Respir Crit Care Med. 2004 Feb 1;169(3):361-6. doi: 10.1164/rccm.200306-752OC. Epub 2003 Nov 3. PMID 14597482
- [Background] De Vito A, Carrasco Llatas M, Vanni A, Bosi M, Braghiroli A, Campanini A, de Vries N, Hamans E, Hohenhorst W, Kotecha BT, Maurer J, Montevecchi F, Piccin O, Sorrenti G, Vanderveken OM, Vicini C. European position paper on drug-induced sedation endoscopy (DISE). Sleep Breath. 2014 Sep;18(3):453-65. doi: 10.1007/s11325-014-0989-6. Epub 2014 May 26. PMID 24859484
- [Background] Aktas O, Erdur O, Cirik AA, Kayhan FT. The role of drug-induced sleep endoscopy in surgical planning for obstructive sleep apnea syndrome. Eur Arch Otorhinolaryngol. 2015 Aug;272(8):2039-43. doi: 10.1007/s00405-014-3162-8. Epub 2014 Jun 28. PMID 24972543
- [Background] Ehsan Z, Mahmoud M, Shott SR, Amin RS, Ishman SL. The effects of anesthesia and opioids on the upper airway: A systematic review. Laryngoscope. 2016 Jan;126(1):270-84. doi: 10.1002/lary.25399. Epub 2015 Jul 21. PMID 26198715
- [Background] Lo YL, Ni YL, Wang TY, Lin TY, Li HY, White DP, Lin JR, Kuo HP. Bispectral Index in Evaluating Effects of Sedation Depth on Drug-Induced Sleep Endoscopy. J Clin Sleep Med. 2015 Sep 15;11(9):1011-20. doi: 10.5664/jcsm.5016. PMID 25979098
- [Background] Hong SD, Dhong HJ, Kim HY, Sohn JH, Jung YG, Chung SK, Park JY, Kim JK. Change of obstruction level during drug-induced sleep endoscopy according to sedation depth in obstructive sleep apnea. Laryngoscope. 2013 Nov;123(11):2896-9. doi: 10.1002/lary.24045. Epub 2013 Aug 5. PMID 23918761
- [Background] Stierer TL, Ishman SL. Bispectral Index in Evaluating Effects of Sedation Depth on Drug-Induced Sleep Endoscopy: DISE or No Dice. J Clin Sleep Med. 2015 Sep 15;11(9):965-6. doi: 10.5664/jcsm.5002. No abstract available. PMID 26285116
- [Background] Chen X, Tang J, White PF, Wender RH, Ma H, Sloninsky A, Kariger R. A comparison of patient state index and bispectral index values during the perioperative period. Anesth Analg. 2002 Dec;95(6):1669-74, table of contents. doi: 10.1097/00000539-200212000-00036. PMID 12456436
- [Background] Schneider G, Mappes A, Neissendorfer T, Schabacker M, Kuppe H, Kochs E. EEG-based indices of anaesthesia: correlation between bispectral index and patient state index? Eur J Anaesthesiol. 2004 Jan;21(1):6-12. doi: 10.1017/s0265021504001024. PMID 14768917
- [Background] Drover D, Ortega HR. Patient state index. Best Pract Res Clin Anaesthesiol. 2006 Mar;20(1):121-8. doi: 10.1016/j.bpa.2005.07.008. PMID 16634419
- [Background] Drover DR, Lemmens HJ, Pierce ET, Plourde G, Loyd G, Ornstein E, Prichep LS, Chabot RJ, Gugino L. Patient State Index: titration of delivery and recovery from propofol, alfentanil, and nitrous oxide anesthesia. Anesthesiology. 2002 Jul;97(1):82-9. doi: 10.1097/00000542-200207000-00012. PMID 12131107
- [Background] Prichep LS, Gugino LD, John ER, Chabot RJ, Howard B, Merkin H, Tom ML, Wolter S, Rausch L, Kox WJ. The Patient State Index as an indicator of the level of hypnosis under general anaesthesia. Br J Anaesth. 2004 Mar;92(3):393-9. doi: 10.1093/bja/aeh082. Epub 2004 Jan 22. PMID 14742326
- [Background] Akhan G, Ayik S, Songu M. Cerebral oxygenation during sleep in patients with obstructive sleep apnea: a near-infrared spectroscopy study. J Otolaryngol Head Neck Surg. 2012 Dec;41(6):437-42. PMID 23700590
- [Background] Pizza F, Biallas M, Wolf M, Werth E, Bassetti CL. Nocturnal cerebral hemodynamics in snorers and in patients with obstructive sleep apnea: a near-infrared spectroscopy study. Sleep. 2010 Feb;33(2):205-10. doi: 10.1093/sleep/33.2.205. PMID 20175404
- [Background] Olopade CO, Mensah E, Gupta R, Huo D, Picchietti DL, Gratton E, Michalos A. Noninvasive determination of brain tissue oxygenation during sleep in obstructive sleep apnea: a near-infrared spectroscopic approach. Sleep. 2007 Dec;30(12):1747-55. doi: 10.1093/sleep/30.12.1747. PMID 18246984
- [Background] Rimpila V, Saaresranta T, Huhtala H, Virkki A, Salminen AV, Polo O. Transcutaneous CO(2) plateau as set-point for respiratory drive during upper airway flow-limitation. Respir Physiol Neurobiol. 2014 Jan 15;191:44-51. doi: 10.1016/j.resp.2013.10.014. Epub 2013 Nov 4. PMID 24200642
- [Background] Carratu P, Ventura VA, Maniscalco M, Dragonieri S, Berardi S, Ria R, Quaranta VN, Vacca A, Devito F, Ciccone MM, Phillips BA, Resta O. Echocardiographic findings and plasma endothelin-1 levels in obese patients with and without obstructive sleep apnea. Sleep Breath. 2016 May;20(2):613-9. doi: 10.1007/s11325-015-1260-5. Epub 2015 Sep 18. PMID 26385777
- [Background] Imai Y, Tanaka N, Usui Y, Takahashi N, Kurohane S, Takei Y, Takata Y, Yamashina A. Severe obstructive sleep apnea increases left atrial volume independently of left ventricular diastolic impairment. Sleep Breath. 2015 Dec;19(4):1249-55. doi: 10.1007/s11325-015-1153-7. Epub 2015 Mar 17. PMID 25778947
- [Background] Wachter R, Luthje L, Klemmstein D, Luers C, Stahrenberg R, Edelmann F, Holzendorf V, Hasenfuss G, Andreas S, Pieske B. Impact of obstructive sleep apnoea on diastolic function. Eur Respir J. 2013 Feb;41(2):376-83. doi: 10.1183/09031936.00218211. Epub 2012 Jul 12. PMID 22790918
- [Background] Hammerstingl C, Schueler R, Wiesen M, Momcilovic D, Pabst S, Nickenig G, Skowasch D. Impact of untreated obstructive sleep apnea on left and right ventricular myocardial function and effects of CPAP therapy. PLoS One. 2013 Oct 11;8(10):e76352. doi: 10.1371/journal.pone.0076352. eCollection 2013. PMID 24146857
- [Background] Tugcu A, Guzel D, Yildirimturk O, Aytekin S. Evaluation of right ventricular systolic and diastolic function in patients with newly diagnosed obstructive sleep apnea syndrome without hypertension. Cardiology. 2009;113(3):184-92. doi: 10.1159/000193146. Epub 2009 Jan 19. PMID 19151552
- [Background] Aydin M, Altin R, Ozeren A, Kart L, Bilge M, Unalacak M. Cardiac autonomic activity in obstructive sleep apnea: time-dependent and spectral analysis of heart rate variability using 24-hour Holter electrocardiograms. Tex Heart Inst J. 2004;31(2):132-6. PMID 15212122
- [Background] Yang A, Schafer H, Manka R, Andrie R, Schwab JO, Lewalter T, Luderitz B, Tasci S. Influence of obstructive sleep apnea on heart rate turbulence. Basic Res Cardiol. 2005 Sep;100(5):439-45. doi: 10.1007/s00395-005-0536-5. Epub 2005 Jun 10. PMID 15944808
- [Background] Zhu K, Chemla D, Roisman G, Mao W, Bazizi S, Lefevre A, Escourrou P. Overnight heart rate variability in patients with obstructive sleep apnoea: a time and frequency domain study. Clin Exp Pharmacol Physiol. 2012 Nov;39(11):901-8. doi: 10.1111/1440-1681.12012. PMID 23006023
- [Background] Kezirian EJ, Hohenhorst W, de Vries N. Drug-induced sleep endoscopy: the VOTE classification. Eur Arch Otorhinolaryngol. 2011 Aug;268(8):1233-1236. doi: 10.1007/s00405-011-1633-8. Epub 2011 May 26. PMID 21614467